CLINICAL TRIAL: NCT01536028
Title: A Double-blind, Randomised, Four-Period Crossover Trial Comparing the Pharmacodynamics and Pharmacokinetics After Single Dose of Biphasic Insulin Aspart 30, Biphasic Insulin Aspart 50, Biphasic Insulin Aspart 70 and Insulin Aspart in Subjects With Type 1 Diabetes
Brief Title: Comparison of the Pharmacodynamics and Pharmacokinetics of Biphasic Insulin Aspart 30, 50, 70 and Insulin Aspart in Subjects With Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: BIASP-1746; 2005-004965-40 (EudraCT Number)
Record Dates: First submitted 2012-02-15; First posted 2012-02-20 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — insulin aspart, insulin aspart protamine drug combination 30:70; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- BIAsp 30 (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70; Drug: insulin aspart
- BIAsp 50 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70; Drug: insulin aspart
- BIAsp 70 (Experimental)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70; Drug: insulin aspart
- IAsp (Active Comparator)
  Interventions: Drug: biphasic insulin aspart 30; Drug: biphasic insulin aspart 50; Drug: biphasic insulin aspart 70; Drug: insulin aspart

INTERVENTIONS:
Drug: biphasic insulin aspart 30 — A single dose administrated subcutaneously (s.c., under the skin) on four separate dosing visits in random order with a washout of 1-2 weeks in-between
Drug: biphasic insulin aspart 50 — A single dose administrated subcutaneously (s.c., under the skin) on four separate dosing visits in random order with a washout of 1-2 weeks in-between
Drug: biphasic insulin aspart 70 — A single dose administrated subcutaneously (s.c., under the skin) on four separate dosing visits in random order with a washout of 1-2 weeks in-between
Drug: insulin aspart — A single dose administrated subcutaneously (s.c., under the skin) on four separate dosing visits in random order with a washout of 1-2 weeks in-between

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to compare the pharmacodynamics and pharmacokinetics after a single dose of biphasic insulin aspart 30, biphasic insulin aspart 50, biphasic insulin aspart 70 and insulin aspart in subjects with type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for at least 12 months
* Serum C-peptide maximum 0.4 ng/mL
* Current basal bolus treatment with soluble human insulin, insulin lispro, insulin glulisine, NPH insulin, insulin detemir or insulin glargine
* BMI (Body Mass Index) maximum 32 kg/m^2
* HbA1c (glycosylated haemoglobin) maximum 9% based on analysis from central laboratory
* Non-smoker

Exclusion Criteria:

* The receipt of any investigational drug within the last 30 days prior to this trial
* Total daily insulin dose at least 1.8 U/kg/day
* Current treatment with IAsp (insulin aspart) products
* A history of drug or alcohol abuse within the last 5 years
* Impaired hepatic function
* Impaired renal function
* Cardiac problems
* Severe, uncontrolled hypertension

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2006-04; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Area under the GIR (glucose infusion rate)-curves in the first two hours post-dosing

SECONDARY OUTCOMES:
Maximum GIR value
Time to maximum GIR value
Area under the GIR-curves
Maximum drug concentration for insulin aspart (IAsp)
Time to maximum IAsp concentration
Area under the curve of the IAsp profiles
Minimum drug concentration in NEFA (Nonesterified fatty acids)
Time to minimum plasma concentration, NEFA
Area under the curve of the NEFA profiles
Adverse events
Hypoglycaemic episodes

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Neuss, Germany

REFERENCES:
- [Result] Heise T, Eckers U, Kanc K, Nielsen JN, Nosek L. The pharmacokinetic and pharmacodynamic properties of different formulations of biphasic insulin aspart: a randomized, glucose clamp, crossover study. Diabetes Technol Ther. 2008 Dec;10(6):479-85. doi: 10.1089/dia.2008.0019. PMID 19049377
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com